CLINICAL TRIAL: NCT04726332
Title: A Dose Escalation and Expansion Study of the Safety and Pharmacokinetics of XL102 as Single-Agent and Combination Therapy in Subjects With Inoperable Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of XL102 as Single-Agent and Combination Therapy in Subjects With Solid Tumors (QUARTZ-101)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL102-101
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Neoplasm Malignant; Epithelial Ovarian Cancer; Triple Negative Breast Cancer; Hormone Receptor Positive Breast Carcinoma; Metastatic Castration-resistant Prostate Cancer
Keywords: cdk7 inhibitor
MeSH Terms: conditions — Neoplasms; Carcinoma, Ovarian Epithelial; Triple Negative Breast Neoplasms | interventions — Fulvestrant; abiraterone; Prednisone

STUDY DESIGN:
Intervention Model Description: Single-agent and combination therapy dose-escalation followed by cohort-expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- XL102 Single-Agent Dose-Escalation Cohorts (Experimental): Subjects will be separated into three separate groups of cohorts. Formulation A consists of: Fasted, with approximately 9 cohorts (A-FC) starting at 20 mg (qd and/or bid) of XL102, Food-Effect Dose-Escalation at 40 mg qd of XL102, with approximately 3 cohorts (A-FE) and Non-Fasted, with approximately 6 cohorts (A-NF).
  Formulation B consists of additional cohorts: Fasted (A-FCFB) starting at 40 mg (qd and/or bid) of XL102 and Non-Fasted (A-NFCFB).
  The dose of the remaining A-FE cohorts will be determined by the Cohort Review Committee (CRC) as well as that of the A-NF, and A-NFCFB cohorts.
  Interventions: Drug: XL102
- XL102 Single-Agent Expansion Cohorts (Experimental): The Maximum Tolerated Dose (MTD) or recommended dose from the dose-escalation stage may be further explored in subjects with triple-negative breast cancer (TNBC) (Cohort D), epithelial ovarian cancer (EOC) (Cohort E), hormone receptor-positive breast cancer (HR+ BC) (Cohort F), and metastatic castration-resistant prostate cancer (mCRPC) (Cohort G).
  Interventions: Drug: XL102
- XL102 + Fulvestrant Dose-Escalation Cohorts (Experimental): Subjects with HR+ BC (Cohort B) will accrue in cohorts of 3-12 subjects in a modified i3+3 design.
  Interventions: Drug: XL102; Drug: Fulvestrant
- XL102 + Abiraterone/Prednisone Dose-Escalation Cohorts (Experimental): Subjects with mCRPC (Cohort C) will accrue in cohorts of 3-12 subjects in a modified i3+3 design.
  Interventions: Drug: XL102; Drug: Abiraterone; Drug: Prednisone
- XL102 + Fulvestrant Expansion Cohorts (Experimental): The MTD or recommended dose from the dose-escalation stage may be further explored in subjects with HR+ BC (Cohort H).
  Interventions: Drug: XL102; Drug: Fulvestrant
- XL102 + Abiraterone/Prednisone Expansion Cohorts (Experimental): The MTD or recommended dose from the dose-escalation stage may be further explored in subjects with mCRPC (Cohort I).
  Interventions: Drug: XL102; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: XL102 — oral doses of XL102
Drug: Fulvestrant — fulvestrant 500 mg administered as an intramuscular (IM) injection every 2 weeks for the first 3 doses and then every 4 weeks.
  Arms: XL102 + Fulvestrant Dose-Escalation Cohorts; XL102 + Fulvestrant Expansion Cohorts
Drug: Abiraterone — abiraterone 1000 mg administered orally once daily.
  Arms: XL102 + Abiraterone/Prednisone Dose-Escalation Cohorts; XL102 + Abiraterone/Prednisone Expansion Cohorts
Drug: Prednisone — prednisone 5 mg administered orally twice daily.
  Arms: XL102 + Abiraterone/Prednisone Dose-Escalation Cohorts; XL102 + Abiraterone/Prednisone Expansion Cohorts

SUMMARY:
This is a Phase 1, open-label, dose-escalation and expansion study evaluating the safety, tolerability, PK, antitumor activity, and effect on biomarkers of XL102 administered orally alone and in multiple combination regimens to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically and radiologically confirmed solid tumor that is inoperable, locally advanced, metastatic, or recurrent.
* Dose-Escalation Stage Cohort A (Solid Tumors): The subject has a solid tumor that is unresectable or metastatic and for which life-prolonging measures do not exist or available therapies are intolerable or no longer effective.
* Dose-Escalation Stage Cohort B and Cohort-Expansion Stage Cohorts F and H (Hormone Receptor-Positive Breast Cancer): Subjects with breast cancer that is hormone receptor-positive (estrogen receptor positive [ER+] and/or progesterone receptor positive [PR+]) and negative for human epidermal growth factor receptor 2 (HER-2 negative [HER-2-]) and who have documented radiographic disease progression during or following their last systemic anticancer therapy for inoperable locally advanced or metastatic disease.
* Dose-Escalation Stage Cohort C and Cohort-Expansion Stage Cohorts G and I (Metastatic Castration-Resistant Prostate Cancer): Subjects with adenocarcinoma of the prostate. Note: Neuroendocrine differentiation and other histological features are permitted if adenocarcinoma is the primary histology.
* Cohort-Expansion Stage Cohort D (Triple Negative Breast Cancer): Subjects with breast cancer that is negative for HER-2, estrogen receptors, and progesterone receptors, and who have documented radiographic disease progression during or following their last systemic anticancer therapy for inoperable locally advanced or metastatic disease.
* Cohort-Expansion Stage Cohort E (Epithelial Ovarian Cancer): Subjects with epithelial ovarian cancer, including primary peritoneal cancer (PPC) and fallopian tube cancer (FTC) who have platinum-resistant disease following treatment with a platinum-containing chemotherapy. Ovarian borderline epithelial tumors (low malignant potential) are excluded.
* Expansion Cohorts: Subjects must have measurable disease per RECIST 1.1 as determined by the Investigator.
* Tumor tissue material (archival or fresh tumor tissue [if it can be safely obtained]).
* Recovery to baseline or ≤ Grade 1 severity (Common Terminology Criteria for Adverse Events version 5 [CTCAE v5]) from AEs, unless AEs are clinically nonsignificant (eg, alopecia) or stable (eg, peripheral neuropathy).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ and marrow function.
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception.
* Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

* Receipt of XL102 or any other selective CDK7 inhibitor.
* Receipt of any cytotoxic chemotherapy therapy or anticancer antibody therapy within 21 days before first dose of study treatment.
* Receipt of any type of small molecule kinase inhibitor within 2 weeks before first dose of study treatment.
* Receipt of any anticancer hormonal therapy within 2 weeks or within 5 half-lives of the agent, whichever is shorter, before first dose of study treatment. HR+BC subjects enrolled in the Combination Cohorts B and H receiving fulvestrant prior to first dose of study treatment are allowed to continue with their fulvestrant treatment. Metastatic CRPC subjects enrolled in the Combination Cohorts C and I receiving abiraterone prior to first dose of study treatment are allowed to continue with their abiraterone treatment.
* Radiation therapy within 14 days before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Known brain tumors and metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.
* Use of strong inhibitors or inducers of cytochrome P450 (CYP) 3A4, and inhibitors of P-glycoprotein (P-gp) or breast cancer resistance protein (BCRP) transporter within 5 half-lives or 4 weeks prior to first dose of study treatment, whichever is shorter.
* Use of a sensitive substrate of CYP3A4, CYP2B6, CYP2C8, CYP2C9, or BCRP transporter within 5 half-lives or 4 weeks prior to first dose of study treatment, whichever is shorter. For subjects with mCRPC in receiving combination treatment with XL102 and abiraterone plus prednisone, use of a substrate of CYP2D6 with a narrow therapeutic index within 5 half-lives or 4 weeks prior to first dose of study treatment, whichever is shorter, is prohibited.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  1. Cardiovascular disorders: i. congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias (eg, ventricular flutter, ventricular fibrillation, torsades de pointes). ii. uncontrolled hypertension defined as sustained blood pressure > 150 mmHg systolic or >90 mm Hg diastolic despite optimal antihypertensive treatment. iii. stroke (including transient ischemic attack [TIA]), myocardial infarction, or other ischemic event or pulmonary embolism (PE) within 6 months before first dose. Note: Subjects with a diagnosis of deep vein thrombosis (DVT) within 6 months before first dose are allowed if managed adequately with anticoagulants and asymptomatic at the time of first dose.
  2. history of any lower gastrointestinal (GI) disorder (such as inflammatory bowel disease [IBD]) or any form of colitis (such as ulcerative colitis or Crohn's disease).
  3. history of upper gastrointestinal (GI) inflammatory disorder (eg, esophagitis, gastritis, or duodenitis), gastroparesis, symptomatic gastroesophageal reflux disease (GERD) despite medical therapy, or gastric or duodenal ulcers within 6 months.
  4. history of major surgical resection involving the stomach or small bowel or any other reason for a malabsorption syndrome.
  5. history of significant bleeding (eg, GI hemorrhage) within 12 weeks before first dose.
  6. active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, acute or chronic hepatitis B or C infection, or a known positive test for tuberculosis infection if supported by clinical or radiographic evidence of disease. Prophylactic use of antibiotics is allowed.
  7. History of COVID-19 unless the subject has clinically recovered from the infection: at least 10 days prior to first dose or sooner, if COVID-19 PCR negative.
  8. moderate to severe hepatic impairment (child-pugh B or C)
  9. requirement for hemodialysis or peritoneal dialysis
  10. history of solid organ, autologous or allogenic stem cell transplant
* Concomitant use of certain medications.
* Uncontrolled, significant intercurrent or recent illness.
* Major surgery within 4 week before first dose of treatment. Minor surgery within 7 days before first dose of treatment. Complete wound healing from surgery must have occurred before first dose of treatment.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms per electrocardiogram (ECG).
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Inability to swallow oral study treatment formulation
* Previously identified allergy or hypersensitivity to study treatment formulation
* Pregnant or lactating females.
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.
* For subjects in Food-Effect Cohorts (A-FE) only: i. Known inability to tolerate high-fat meal provided on Day 1 ii. Allergy to meal components or dietary restrictions iii. Unable to fast for 4 hours predose and 2 hours post dose on Day 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Dose-Escalation Stage: MTD/recommended dose for XL102 | Approximately 18 months
  To determine the MTD and/or RD for further evaluation of XL102 when administered orally alone and in combination therapy in subjects with advanced solid tumors
Cohort-Expansion Stage: Objective Response Rate (ORR) | Approximately 12 months
  To evaluate preliminary efficacy of XL102 when administered alone and in combination therapy by estimating the ORR as assessed by the Investigator per RECIST 1.1

SECONDARY OUTCOMES:
Safety of XL102 as evaluated by Incidence and Severity of Adverse Events (AEs) | Approximately 30 months
  To evaluate the safety of XL102 when administered orally alone and in combination therapy through the evaluation of overall incidence of AEs, severity grade, relationship to study treatment, and laboratory tests.
Tolerability of XL102 as evaluated by Study Treatment Exposure, Dose Intensity and Modifications, and Study Treatment Discontinuation due to AE | Approximately 30 months
  To evaluate the tolerability of XL102 when administered orally alone and in combination therapy through the evaluation of study treatment exposure, dose intensity, dose modifications, and study treatment discontinuation due to AE.
Dose-Escalation Stage: Drug-Drug Interactions | Approximately 18 months
  To assess drug-drug interactions between XL102 and combination agents
Dose-Escalation Stage: Time to Maximum Plasma Concentration (Tmax) | Approximately 18 months
  To evaluate the Tmax of XL102 alone and in combination therapy
Dose-Escalation Stage: Maximum Plasma Concentration (Cmax) | Approximately 18 months
  To evaluate the Cmax of XL102 alone and in combination therapy
Dose-Escalation Stage: Area Under the Plasma Concentration-Time Curve Over the Last 24-hour Dosing Interval (AUC 0-24) | Approximately 18 months
  To evaluate the AUC 0-24 of XL102 alone and in combination therapy
Dose-Escalation Stage: Terminal Half-Life | Approximately 18 months
  To evaluate the terminal half-life of XL102 alone and in combination therapy
Dose-Escalation Stage: Apparent Clearance (CL/F) | Approximately 18 months
  To evaluate the CL/F of XL102 alone and in combination therapy

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Exelixis Clinical Site #4, Atlanta, Georgia
  - Exelixis Clinical Site #3, Boston, Massachusetts
  - Exelixis Clinical Site #2, Dallas, Texas
  - Exelixis Clinical Site #5, Houston, Texas
  - Exelixis Clinical Site #1, San Antonio, Texas

REFERENCES:
- [Derived] Gaur T, Poddutoori R, Khare L, Bagal B, Rashmi S, Patkar N, Tembhare P, Pg S, Shetty D, Dutt A, Zhang Q, Konopleva M, Platzbeckar U, Gupta S, Samajdar S, Ramchandra M, Khattry N, Hasan SK. Novel covalent CDK7 inhibitor potently induces apoptosis in acute myeloid leukemia and synergizes with Venetoclax. J Exp Clin Cancer Res. 2023 Jul 29;42(1):186. doi: 10.1186/s13046-023-02750-w. PMID 37507802